CLINICAL TRIAL: NCT06787755
Title: Persistent COVID-19 Symptoms in Minia, Upper Egypt: an Observational Cross-sectional Study
Brief Title: Persistent COVID-19 Symptoms in Minia
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Marwa Kamal Ahmed Tolba, Associate professor, Fayoum University
Other Study IDs: : Persistent COVID-19 symptoms
Record Dates: First submitted 2025-01-19; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: COVID - 19
Keywords: covid19; risk factors; self-medication
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective This study aims to identify the nature and prevalence of persistent symptoms in patients discharged from Minya University hospitals in Egypt after recovery from COVID-19, the severity of these symptoms, and the possible risk factors associated with them.

DETAILED DESCRIPTION:
This is a cross-sectional observational retrospective study. The study population included patients, both hospitalized and non-hospitalized, who were diagnosed with COVID-19. Demographic information, symptom severity, present comorbidities, and persistent COVID-19 symptoms were collected. SPSS software was used for the statistical analysis, and p-values less than 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria Patients were included in this study if they tested positive for COVID-19 at the time of their illness (positive COVID-19 polymerase chain reaction [PCR] test) or if laboratory, clinical, and radiological criteria suggested the infection with COVID-19, and the severity of their symptoms ranged from asymptomatic to severe. Both hospitalized and non-hospitalized patients were included.

Exclusion Criteria:

Exclusion criteria Patients excluded were frail or at the end of their life or had severe cognitive dysfunction, as well as patients <18 years of age.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional observational retrospective survey study in which we collected information about any persistent or new symptoms after recovery from COVID-19. The average time after recovery from COVID was 6 months at the time of patient interviews, and the median duration of symptoms was 14 days. We collected various patient data including their medical history before COVID-19, treatments they received during their illness, and self-reported use of unprescribed antibiotics in home-isolated patients.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Long COVID-19 has been an increasingly prevalent concern in the medical community for the last two years and is still a burden on the healthcare system worldwide | 2years
  Constitutional and neurological manifestations are two of the most persistent symptoms. Lack of appropriate levels of awareness about long COVID-19, as well as the tendency of patients in this demographic to self-medicate are leading causes of the underreporting of long COVID-19 symptoms in this region

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa, Al Fayyum, Egypt

REFERENCES:
- [Result] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937